CLINICAL TRIAL: NCT01643044
Title: Computer-delivered SBIRT for Alcohol Use in Pregnancy: Planning a Stage II Trial
Brief Title: Computer-delivered Screening and Brief Intervention for Alcohol Use in Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R34AA020056 (NIH); R34AA020056 (NIH)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Alcohol Abuse
Keywords: pregnancy; screening; motivation
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol intervention (Experimental): Participants in this condition review tailored videos and normed feedback regarding their alcohol use and possible consequences of drinking. Next participants view a goal setting section describing possible ways to quit drinking alcohol and the participant is able to indicate a change goal (if any) and is helped through a specific change plan, should they set a change goal.
  Interventions: Behavioral: Computer-delivered, brief intervention on alcohol use
- Control (Placebo Comparator): Participants randomized into the control condition complete assessment and a time-matched interactive session on infant nutrition.
  Interventions: Behavioral: Nutrition time control/placebo intervention

INTERVENTIONS:
Behavioral: Nutrition time control/placebo intervention — This time-control intervention, designed in part to help promote research assistant blinding as to participant condition, focused on proper infant nutrition using a computer-delivered, interactive format and videos.
  Arms: Control
Behavioral: Computer-delivered, brief intervention on alcohol use — A single 20-minute interactive computer-delivered intervention designed to promote motivation to change prenatal alcohol use, without presuming the participant to be currently using alcohol while pregnant.
  Arms: Alcohol intervention

SUMMARY:
The purpose of this study is to lay the ground work for a fully powered clinical trial of a computer-delivered screener and intervention for alcohol use during pregnancy. The pilot study will include:

1. Evaluation of the usefulness of handheld devices and anonymous screening for self report of at-risk alcohol use among pregnant women.
2. Assessing the validity of an alcohol biomarker, Ethyl Glucoronide (EtG), for the detection of at-risk drinking in pregnant women.
3. Evaluation of the efficacy of a computer-delivered brief intervention and use of tailored handouts to supplement the computer-based brief intervention focusing on alcohol use during pregnancy.

DETAILED DESCRIPTION:
Infants born to African-American and/or low SES women appear to be at increased risk of adverse effects due to prenatal exposure to alcohol. Computer-delivered SBIRT approaches may provide consistent screening and evidence-based brief interventions, at low cost, without requiring substantial investments of time or energy from medical staff. However, several Stage I steps are necessary before moving to a Stage II clinical trial. This R34 application will therefore lay the groundwork for a fully powered clinical trial of a computer-delivered SBIRT for alcohol use during pregnancy. It will do so through the conduct of five key preliminary studies, including: (1) evaluation of the utility of handheld mobile devices and an anonymous self-interview format in screening for at-risk drinking among patients attending a prenatal clinic; (2) modification of an existing computer-delivered motivational intervention for alcohol use during pregnancy, to previously set standards of acceptability (to experts as well as representative pregnant women); (3) development of an evidence-based tailored messaging supplement to the single-session brief intervention; (4) examining the validity of, and cut scores for, the biomarker Ethyl Glucoronide (EtG) in pregnant women; and (5) collecting data on the acceptability, feasibility, and estimated effect size of the modified computer-delivered intervention through an N = 50 Phase I randomized clinical trial. Participants in this trial will be a diverse sample of women at-risk for alcohol use during pregnancy, the majority of whom will be African-American and/or low SES. These key preparatory steps will greatly facilitate the subsequent development of an R01 application to conduct a Stage II clinical trial for alcohol use during pregnancy. These steps will also provide important preliminary data on (a) a novel method for risk factor screening in primary care; (b) the potential utility of EtG as a biomarker for alcohol use during pregnancy and in the perinatal period; and (c) the effect size estimate for a fully computer-delivered, combined brief interactive/tailored messaging intervention requiring only a single contact. If successful, this line of research could lead to a highly cost-effective, high-reach intervention for alcohol use during pregnancy; these reductions in alcohol use could in turn have a meaningful population impact on Fetal Alcohol Spectrum Disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* intention to carry pregnancy to term
* self-reported alcohol use
* willingness to be sent tailored messages
* gives consent to access medical records for collection of birth outcome data

Exclusion Criteria:

* unable to communicate in English
* less than 4 months before delivery due date

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alcohol Intervention | Control
Started | 24 | 24
Completed | 20 | 19
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Miscarried baby | 2 | 2
Not completed — Delivered outside of hospital | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alcohol Intervention | Control | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 21 | 39
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Alcohol use will be measured at the time of delivery of their infant by self-report and urine analysis. The number represents the number of participants who were abstinent (reported no alcohol use and had a negative toxicology urine screen) from alcohol for the past 90 days.
Time Frame: self-reported use during 90 days prior to delivery of their baby
Measure: Number; unit: participants
Arm/Group | Alcohol Intervention | Control
Number analyzed (Participants) | 20 | 19
participants | 18 | 14

ADVERSE EVENTS:
Arm/Group | Alcohol Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No